CLINICAL TRIAL: NCT02506010
Title: SpO2 Accuracy Validation of a USB Pulse Oximetry Monitor Interface Cable Via Reference Co-Oximetry
Brief Title: Accuracy Validation of a Pulse Oximetry Monitor
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decided not to run this study.
Sponsor: Medtronic - MITG (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0499
Record Dates: First submitted 2015-07-14; First posted 2015-07-22 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to conduct an oxygen saturation (SpO2) accuracy validation comparing prototype pulse oximeter oxygen saturation measurements directly to arterial blood saturation during non-motion conditions over the range of 60-100% SaO2 as measured by Reference CO-Oximetry. Additionally, the prototype pulse oximeter pulse rate measurements will be compared to 3-lead ECG heart rate measurements made via a multi-parameter monitor.

DETAILED DESCRIPTION:
The description of this study is to conduct an oxygen saturation (SpO2) accuracy validation comparing prototype pulse oximeter oxygen saturation measurements directly to arterial blood saturation during non-motion conditions over the range of 60-100% SaO2 as measured by Reference CO-Oximetry. Additionally, the prototype pulse oximeter pulse rate measurements will be compared to 3-lead ECG heart rate measurements made via a multi-parameter monitor.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking, or who have refrained from smoking for 2 days
* male or female of any race
* 18-45 years.
* Subjects must have the ability to understand and provide written informed consent as well as be willing to comply with study procedures.
* To be eligible to participate in the study, the subject must clear a recent physical (12-lead ECG, medical history and blood test for sickle cell disease.) prior to enrollment

Exclusion Criteria:

* - morbid obesity (defined as BMI > 39.5),
* injuries, deformities or abnormalities or piercings that may prevent proper application of the device under test, compromised circulation,
* subjects with known respiratory conditions (smokers with COHb levels >3%, flu, pneumonia, bronchitis, shortness of breath/ respiratory distress, severe asthma, emphysema, COPD),
* subjects with known heart or cardiovascular conditions (uncontrolled hypertension, heart arrhythmias other than sinus arrhythmia, previous heart attack, blocked artery, history of myocardial ischemia, angina, myocardial infarction, congestive heart failure or cardiomyopathy, history of stroke, transient ischemic attack or carotid artery disease),
* other known health condition (diabetes, thyroid disease, kidney disease / chronic renal impairment, history of seizures (except childhood febrile seizures) or epilepsy, or unexplained syncope, recent history of frequent migraine headaches, recent head injury, cancer / chemotherapy
* women actively trying to get pregnant or are pregnant,
* clotting disorders (history of bleeding disorders or current use of blood thinners, Hemophilia, blood clots)
* Sickle cell disease
* Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
* Unwillingness or inability to remove colored nail polish or artificial nails from test digit(s)
* Prior or known allergies to: lidocaine (or similar pharmacological agents, e.g., Novocain) or heparin
* Recent arterial cannulation (i.e., less than 30 days prior to study date), Six or more arterial cannulations of each (right & left) radial artery, history of clinically significant complications from previous arterial cannulation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be ten to fifteen male and female subjects of any race, ranging in pigmentation from light to dark to meet the study design requirements
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The OxiCable pulse rate measurement performance is an ARMS of 3 or better over the full range 60-100% SaO2. | 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Ransom, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study was cancelled.